CLINICAL TRIAL: NCT05327179
Title: Effects of Action Observation Therapy and Video-Based Play Therapy on the Upper Extremity and Trunk in Children With Unilateral Cerebral Palsy in the Framework of the International Classification of Functioning, Disability, and Health
Brief Title: Effects of Action Observation Therapy and Video-Based Play Therapy on Children With Unilateral Cerebral Palsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sinem Erturan (Other)
Responsible Party: Sponsor-Investigator, Sinem Erturan, research assistant, Gazi University
Organization: Gazi University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020 - 698
Record Dates: First submitted 2022-04-07; First posted 2022-04-14 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Cerebral Palsy; Upper Extremity Problem
Keywords: cerebral palsy; upper extremity; virtual rehabilitation; action observation treatment
MeSH Terms: conditions — Cerebral Palsy | interventions — Telerehabilitation

STUDY DESIGN:
Intervention Model Description: Individual with cerebral palsy will be assigned to group 1 or group 2 by simple randomization using the "Research Randomiser" program (http://www.randomizer.org/) prior to treatment.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Action Observation Treatment
  Interventions: Other: Action Observation Treatment
- Group 2 (Experimental): Virtual Rehabilitation
  Interventions: Other: Virtual Rehabilitation

INTERVENTIONS:
Other: Action Observation Treatment — Action Observation Treatment program will be applied to the group 1 for 3 weeks, 5 days a week, 30 minutes a day. In the videos prepared, activities including daily life activities for the wrist, elbow and shoulder (emptying water from the glass, throwing sugar into the glass, painting, using clothespins, spoons, etc.) will be included.
  Arms: Group 1
Other: Virtual Rehabilitation — Virtual Rehabilitation program will be applied to the group 2 for 3 weeks, 5 days a week, 30 minutes a day. Among the games, games that will improve daily life activities for the wrist, elbow and shoulder (steering wheel, popping balloons, touching the aquarium, etc.) will be selected.
  Arms: Group 2

SUMMARY:
Cerebral Palsy (CP) defines a group of permanent disorders in the development of movement and posture, which occur in the developing fetal and newborn brain, due to non-progressive disorders, leading to activity limitations. In addition to the traditional rehabilitation interventions used in upper extremity rehabilitation, a new treatment method, Action Observation Therapy (AOT), has been added recently with the discovery of the Mirror Neuron System. AOT; By watching the videos prepared, mirror neurons are activated and these activities are learned through imitation. Activation of mirror neurons strengthens voluntary motor movement by strengthening the affected nerve pathways or by creating alternative pathways. AOT is an easily applicable method as telerehabilitation because it is based on watching and replaying video recordings. Virtual Rehabilitation (VR); It is another treatment approach applied to improve the motor functions of children with CP and created with the contribution of developing technology. It has been reported that activities have a positive effect on motor learning due to their intense, task-oriented, active participation and high motivation. Within the scope of this thesis, the effect of AOT and VR to be applied at home, which has been on the agenda for upper extremity, on the trunk and upper extremity will be examined in detail and a contribution will be made to the literature.

DETAILED DESCRIPTION:
Cerebral Palsy (CP) defines a group of permanent disorders in the development of movement and posture that occur in the developing fetal and newborn brain, due to non-progressive disorders, leading to activity limitations. Unilateral CP (uCP) accounts for 38% of cases. These children complain of motor and sensory disorders that are more prominent on one side of the body, usually in the upper extremity (UE). These sensorimotor disorders typically limit their ability to perform activities of daily living, negatively affecting participation and quality of life. Therefore, in the last ten years, research on UE interventions for children with uCP has been focused on; While trying to develop existing methods, new treatment methods are tried to be created. There are various treatment modalities that aim to relieve UE function disorders and reduce activity limitations. It is very important to determine the most effective treatment method. However, there are few randomized controlled studies measuring clinical outcomes in children with uCP. New intervention strategies based on sound methodological and scientific foundations are needed.

It has been reported that motor learning is the basis of UE treatments applied in CP and reported to be effective. Based on neurophysiological findings, there are studies suggesting that AOT and VR treatment approaches accelerate the motor learning process. AOT; It includes observing selected UE actions and actively imitating the observed action. AOT has been previously used in the treatment of upper extremity in patients with chronic stroke, recovery of frostbite phenomenon in Parkinson's disease, treatment of lower and upper extremities in pediatric rehabilitation, and recovery of limb function after orthopedic surgery and has been reported in studies. Recent studies, especially in children with uCP, have reported promising results. In general, telerehabilitation is an effective, flexible, personalized and relatively cost-effective intervention, which strengthens the hypothesis that home rehabilitation services are a viable alternative to routine care. AOT can be easily performed at home as it is an approach based on careful observation and active imitation of actions. approach has been reported. Studies have reported that VR improves posture, balance, upper extremity function, and trunk control. There is no study in the literature examining the effects of motor learning-based AOT and VR applied at home on UE and body within the framework of international functionality, disability and health classification. Within the scope of the study, a contribution will be made to the literature, which has been reported to be insufficient in studies on UE treatments.

ELIGIBILITY:
Inclusion Criteria:

* The clinical type is spastic hemiparetic CP.
* Upper extremity spasticity value between 0 and 3 according to Modified Ashworth.
* To have the cognitive level to understand simple instructions.
* It is largely the absence of auditory and visual loss.

Exclusion Criteria:

* Not volunteering to participate in the study.

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2022-10-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Sociodemographic Data Form | Before starting treatment
  Information such as gender, age, clinical type, extremity involvement, dominant extremity, birth weight, assistive devices used of the cases will be recorded in the prepared sociodemographic data form
Joint Range of Motion (ROM) Measurement | Before starting treatment
  Individuals' ROM degrees will be evaluated before and after the treatment using a universal goniometer in the supine position. Individuals' shoulder flexion, abduction, internal and external rotation, elbow and wrist flexion and extension painless active ROM measurements will be evaluated and recorded bilaterally.
Pediatric Quality of Life Inventory | Before starting treatment
  The Pediatric Quality of Life Inventory (PedsQL™) is a modular instrument for measuring health-related quality of life dimensions in children and adolescents ages 2-18 years. The PedsQL™ 4.0 Generic Core Scales are multidimensional (physical, emotional, social, school/role functioning) child self-report and parent proxy report scales developed as a generic measure to be integrated with the PedsQL™ disease-specific modules.
The Jebsen Hand Function Test | Before starting treatment
  The Jebsen Hand Function Test (JHFT) was developed to provide a standardized and objective evaluation of fine and gross motor hand function using simulated activities of daily living. It has 7 items and takes approximately 15-45 minutes to administer.
  Item 1: Writing, Item 2: Card Turning, Item 3: Small Common Objects, Item 4: Simulated feeding, Item 5: Checkers, Item 6: Large Light Object, Item 7: Large Heavy Objects
ABILHAND-Kids | Before starting treatment
  ABILHAND-Kids is a measure of manual ability for children with upper limb impairments. The scale measures a person's ability to manage daily activities that require the use of the upper limbs, whatever the strategies involved. The ABILHAND-Kids questionnaire assesses manual ability as a test focused on the child's difficulty perceived by the child's parents.
  The questionnaire was developed using the Rasch measurement model which provides a method to convert the raw scores into a linear measure located on a unidimensional scale.
  ABILHAND-Kids has been calibrated in children with cerebral palsy according to the difficulty of children in performing manual activities as perceived by their parents.
The Quality of Upper Extremity Skills Test | Before starting treatment
  The Quality of Upper Extremity Skills Test is an outcome measure designed to evaluate movement patterns and hand function in children with cerebral palsy. The QUEST is both reliable and valid. There are 36 items that evaluate dissociated movements, grip, protective extension, and weight bearing
Selective Control of the Upper Extremity Scale | Before starting treatment
  This test was developed to evaluate the selective motor control of the upper extremity. It is a very practical and useful video-based assessment tool that can be applied in less than 15 minutes. No special equipment is required other than a video camera. It offers the opportunity to evaluate the selective movements of the shoulder, elbow, forearm, wrist and fingers for both right and left extremities. The person administering the test passively shows the participant the movements they are asked to do. Then the participant is asked to actively perform the movement shown. While performing the participant movements; Head, trunk and other extremity movements are taken with a video camera to provide the opportunity to observe. The degree of selective motor control is determined as 0-3 points for each joint, depending on the person's ability to perform movements and their shape.
Trunk Control Measurement Scale | Before starting treatment
  The Trunk Control Measurement Scale (TCMS) was used to evaluate the trunk control of the individuals participating in the study. The TCMS includes 15 items that measure static and dynamic sitting balance, the two main components of trunk control. The Static Sitting Balance Scale (item 1-5) evaluates the ability to maintain a stable trunk posture during movements of the upper and lower extremities. The Dynamic Sitting Balance Scale (item 6-15) is divided into two subscales, the selective movement control scale and the dynamic reaching scale. The total score is between 0-58. A higher score indicates better performance.
Gross grip strength | Before starting treatment
  The Association of American Handheld Runners (AAHR) set a standard position to measure hand grip strength. According to the standard position; The patient will be in a sitting position, shoulders in adduction, elbows in 90 degrees flexion, and forearm and wrist in neutral position. The unit of grip force will be accepted as Newton.
Pinch force | Before starting treatment
  Pinch force was evaluated using a pinchmeter. In cases; Type, lateral and triple grip measurements will be made. The measurement position is recommended by the American Association of Hand Therapists; the shoulder will be in adduction and rotation-neutral position, the elbow will be in 90-degree flexion, and the forearm and wrist will be in neutral position. These conditions will be provided while the patient is in a sitting position.
Childhood Health Assessment Questionaire | Before starting treatment
  CHAQ; It consists of 8 subsections and 30 questions: dressing and personal care, standing up, eating, walking, body care, reaching, holding, activities. In addition, the use of assistive devices, devices, pain and well-being are questioned. A separate and total score is calculated for each subsection. Each question is evaluated as no difficulty: 3, with some difficulty: 2, with great difficulty: 1, unable to do: 0 points. In our study, the cases in both groups will be evaluated with CHAQ.
Sociodemographic Data Form | After 3 weeks of treatment (treatment is 15 sessions)
  Information such as gender, age, clinical type, extremity involvement, dominant extremity, birth weight, assistive devices used of the cases will be recorded in the prepared sociodemographic data form
Joint Range of Motion (ROM) Measurement | After 3 weeks of treatment (treatment is 15 sessions)
  Individuals' ROM degrees will be evaluated before and after the treatment using a universal goniometer in the supine position. Individuals' shoulder flexion, abduction, internal and external rotation, elbow and wrist flexion and extension painless active ROM measurements will be evaluated and recorded bilaterally.
Pediatric Quality of Life Inventory | After 3 weeks of treatment (treatment is 15 sessions)
  The Pediatric Quality of Life Inventory (PedsQL™) is a modular instrument for measuring health-related quality of life dimensions in children and adolescents ages 2-18 years. The PedsQL™ 4.0 Generic Core Scales are multidimensional (physical, emotional, social, school/role functioning) child self-report and parent proxy report scales developed as a generic measure to be integrated with the PedsQL™ disease-specific modules.
The Jebsen Hand Function Test | After 3 weeks of treatment (treatment is 15 sessions)
  The Jebsen Hand Function Test (JHFT) was developed to provide a standardized and objective evaluation of fine and gross motor hand function using simulated activities of daily living. It has 7 items and takes approximately 15-45 minutes to administer.
  Item 1: Writing, Item 2: Card Turning, Item 3: Small Common Objects, Item 4: Simulated feeding, Item 5: Checkers, Item 6: Large Light Object, Item 7: Large Heavy Objects
ABILHAND-Kids | After 3 weeks of treatment (treatment is 15 sessions)
  ABILHAND-Kids is a measure of manual ability for children with upper limb impairments. The scale measures a person's ability to manage daily activities that require the use of the upper limbs, whatever the strategies involved. The ABILHAND-Kids questionnaire assesses manual ability as a test focused on the child's difficulty perceived by the child's parents.
  The questionnaire was developed using the Rasch measurement model which provides a method to convert the raw scores into a linear measure located on a unidimensional scale.
  ABILHAND-Kids has been calibrated in children with cerebral palsy according to the difficulty of children in performing manual activities as perceived by their parents.
The Quality of Upper Extremity Skills Test | After 3 weeks of treatment (treatment is 15 sessions)
  The Quality of Upper Extremity Skills Test is an outcome measure designed to evaluate movement patterns and hand function in children with cerebral palsy. The QUEST is both reliable and valid. There are 36 items that evaluate dissociated movements, grip, protective extension, and weight bearing
Selective Control of the Upper Extremity Scale | After 3 weeks of treatment (treatment is 15 sessions)
  This test was developed to evaluate the selective motor control of the upper extremity. It is a very practical and useful video-based assessment tool that can be applied in less than 15 minutes. No special equipment is required other than a video camera. It offers the opportunity to evaluate the selective movements of the shoulder, elbow, forearm, wrist and fingers for both right and left extremities. The person administering the test passively shows the participant the movements they are asked to do. Then the participant is asked to actively perform the movement shown. While performing the participant movements; Head, trunk and other extremity movements are taken with a video camera to provide the opportunity to observe. The degree of selective motor control is determined as 0-3 points for each joint, depending on the person's ability to perform movements and their shape.
Trunk Control Measurement Scale | After 3 weeks of treatment (treatment is 15 sessions)
  The Trunk Control Measurement Scale (TCMS) was used to evaluate the trunk control of the individuals participating in the study. The TCMS includes 15 items that measure static and dynamic sitting balance, the two main components of trunk control. The Static Sitting Balance Scale (item 1-5) evaluates the ability to maintain a stable trunk posture during movements of the upper and lower extremities. The Dynamic Sitting Balance Scale (item 6-15) is divided into two subscales, the selective movement control scale and the dynamic reaching scale. The total score is between 0-58. A higher score indicates better performance.
Gross grip strength | After 3 weeks of treatment (treatment is 15 sessions)
  The Association of American Handheld Runners (AAHR) set a standard position to measure hand grip strength. According to the standard position; The patient will be in a sitting position, shoulders in adduction, elbows in 90 degrees flexion, and forearm and wrist in neutral position. The unit of grip force will be accepted as Newton.
Pinch force | After 3 weeks of treatment (treatment is 15 sessions)
  Pinch force was evaluated using a pinchmeter. In cases; Type, lateral and triple grip measurements will be made. The measurement position is recommended by the American Association of Hand Therapists; the shoulder will be in adduction and rotation-neutral position, the elbow will be in 90-degree flexion, and the forearm and wrist will be in neutral position. These conditions will be provided while the patient is in a sitting position.
Childhood Health Assessment Questionaire | After 3 weeks of treatment (treatment is 15 sessions)
  CHAQ; It consists of 8 subsections and 30 questions: dressing and personal care, standing up, eating, walking, body care, reaching, holding, activities. In addition, the use of assistive devices, devices, pain and well-being are questioned. A separate and total score is calculated for each subsection. Each question is evaluated as no difficulty: 3, with some difficulty: 2, with great difficulty: 1, unable to do: 0 points. In our study, the cases in both groups will be evaluated with CHAQ.

CONTACTS AND LOCATIONS:
Overall Officials: sinem erturan, MSc, Principal Investigator — bulentelbasan@gmail.com
Locations (1):
- Gazi University, Ankara, None Selected, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No